CLINICAL TRIAL: NCT04856358
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of GLPG3121-modified Release Formulation in Adult, Healthy, Male Subjects
Brief Title: A Study to Evaluate How Well Single and Multiple Doses of GLPG3121-modified Release Formulation Are Tolerated in Healthy, Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG3121-CL-103; 2020-004174-21 (EudraCT Number)
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part 1 Single Ascending Dose (SAD) and Part 2 Multiple Ascending Dose (MAD) are randomized, double-blind, placebo-controlled; Part 3 Food-effect (FE) is randomized, open-label, crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- GLPG3121 SAD (Experimental): Single doses of GLPG3121 at up to 3 dose levels in ascending order
  Interventions: Drug: GLPG3121
- Placebo SAD (Placebo Comparator): Single doses of placebo
  Interventions: Drug: Placebo
- GLPG3121 MAD (Experimental): Multiple doses of GLPG3121 at up to 3 dose levels in ascending order
  Interventions: Drug: GLPG3121
- Placebo MAD (Placebo Comparator): Multiple doses of placebo
  Interventions: Drug: Placebo
- GLPG3121 FE fed (Experimental): Single dose of GLPG3121 in fed state
  Interventions: Drug: GLPG3121
- GLPG3121 FE fasted (Experimental): Single dose of GLPG3121 in fasted state
  Interventions: Drug: GLPG3121

INTERVENTIONS:
Drug: GLPG3121 — GLPG3121 modified-release tablet
  Arms: GLPG3121 FE fasted; GLPG3121 FE fed; GLPG3121 MAD; GLPG3121 SAD
Drug: Placebo — Matching placebo
  Arms: Placebo MAD; Placebo SAD

SUMMARY:
The aim of the study is to examine the safety and tolerability of GLPG3121-modified release formulation when given to healthy male subjects once as a single dose or multiple times over a period of 14 days in fasting condition or after a standard breakfast.

The study will evaluate how the body absorbs and breaks down GLPG3121, and how GLPG3121 and the major breakdown product of GLPG3121 are eliminated from the body. In addition, the study will investigate the effect of food (high-fat) after a single oral dose of GLPG3121 as modified release tablet.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 55 years of age (extremes included), on the date of signing the informed consent form (ICF).
* A body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests, available at screening and prior to randomization. Hemoglobin, neutrophil, lymphocyte, and platelet counts must be above the lower limit of normal range. Total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), and serum creatinine must be no greater than the upper limit of normal (ULN). Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator.
* Subject must be able and willing to comply with restrictions on prior and concomitant medication.
* Negative screen for drugs (amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, tricyclic antidepressants) and alcohol.

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Known hypersensitivity to investigational product (IP) ingredients or history of a significant allergic reaction to IP ingredients as determined by the investigator.
* Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or history of hepatitis from any cause with the exception of hepatitis A that was resolved at least 3 months prior to first dosing of the IP.
* History of or a current immunosuppressive condition (e.g. human immunodeficiency virus [HIV] infection).
* Having any illness, judged by the investigator as clinically significant, in the 3 months prior to first dosing of the IP.
* Presence or sequelae of gastrointestinal, liver, kidney (estimated glomerular filtration rate [eGFR] <=90 mL/min/1.73 m2, using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.

This list only contains the key exclusion criteria.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment emergent adverse events (TEAEs), treatment-emergent serious adverse events, and TEAEs leading to treatment discontinuations | From screening through study completion, an average of 8 months
  To evaluate the safety and tolerability of single and multiple ascending oral doses of GLPG3121-modified-release formulation (GLPG3121-MR), in adult, healthy, male subjects compared with placebo

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG3121 in SAD | Between Day 1 pre-dose and Day 6
  To evaluate the pharmacokinetics (PK) of single ascending oral doses of GLPG3121 in adult, healthy, male subjects
Cmax of GLPG3121's main metabolite in SAD | Between Day 1 pre-dose and Day 6
  To evaluate the PK of single ascending oral doses of GLPG3121's metabolite in adult, healthy, male subjects
Cmax of GLPG3121 in MAD | Between Day 1 pre-dose and Day 19
  To evaluate the PK of multiple ascending oral doses of GLPG3121 in adult, healthy, male subjects
Cmax of GLPG3121's main metabolite in MAD | Between Day 1 pre-dose and Day 19
  To evaluate the PK of multiple ascending oral doses of GLPG3121's main metabolite in adult, healthy, male subjects
Area under the plasma concentration-time curve (AUC) of GLPG3121 in SAD | Between Day 1 pre-dose and Day 6
  To evaluate the PK of single ascending oral doses of GLPG3121 in adult, healthy, male subjects
AUC of GLPG3121's main metabolite in SAD | Between Day 1 pre-dose and Day 6
  To evaluate the PK of single ascending oral doses of GLPG3121's main metabolite in adult, healthy, male subjects
AUC of GLPG3121 in MAD | Between Day 1 pre-dose and Day 19
  To evaluate the PK of multiple ascending oral doses of GLPG3121 metabolite in adult, healthy, male subjects
AUC of GLPG3121's main metabolite in MAD | Between Day 1 pre-dose and Day 19
  To evaluate the PK of multiple ascending oral doses of GLPG3121's main metabolite in adult, healthy, male subjects
Terminal elimination half-life (t1/2) of GLPG3121 in SAD | Between Day 1 pre-dose and Day 6
  To evaluate the PK of single ascending oral doses of GLPG3121 in adult, healthy, male subjects
t1/2 of GLPG3121's main metabolite in SAD | Between Day 1 pre-dose and Day 6
  To evaluate the PK of single ascending oral doses of GLPG3121's main metabolite in adult, healthy, male subjects
t1/2 of GLPG3121 in MAD | Between Day 1 pre-dose and Day 19
  To evaluate the PK of multiple ascending oral doses of GLPG3121 in adult, healthy, male subjects
t1/2 of GLPG3121's main metabolite in MAD | Between Day 1 pre-dose and Day 19
  To evaluate the PK of multiple ascending oral doses of GLPG3121's main metabolite in adult, healthy, male subjects

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Petkova, MD, Study Director — Galapagos NV
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No